CLINICAL TRIAL: NCT05763511
Title: Improved Diagnosis of Ovarian Cancer by Use of Circulating Tumor DNA as a Biomarker
Status: Recruiting | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Ina Marie Dueholm Hjorth, Medical doctor, PhD student, University of Aarhus
Other Study IDs: Ovarian cancer ctDNA
Record Dates: First submitted 2022-07-04; First posted 2023-03-10 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Ovarian Neoplasms; Ovary Cancer; Ovarian Cysts
MeSH Terms: conditions — Ovarian Neoplasms; Ovarian Cysts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and tumor tissue (after informed consent)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project investigates circulating tumor DNA (ctDNA) in patients with suspected ovarian malignancy.

We hypothesize that measurement of ctDNA in women with suspected ovarian cancer can improve the diagnostic efficiency for preoperative differentiation between benign and malignant masses.

Specifically, we hope to determine the diagnostic efficiency of ctDNA alone and ctDNA in combination with imaging modalities (ultrasonography, MRI, PET-CT) and CA 125 for preoperative differentiation between benign and malignant adnexal masses. Based on this, we hope to develop an improved diagnostic algorithm.

The mutational profile and relation to tumour type, stage, treatment response and prognosis will be explored.

Analyses of blood and tissue samples will be used to examine the disease development and biology.

Blood samples, tumour tissue and data on imaging modalities as well as CA 125 will be collected prospectively in consecutive women referred to Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Suspected ovarian neoplasm
* Informed consent

Exclusion Criteria:

* Inability to give informed consent
* Previous ovarian cancer diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred due to suspected ovarian cancer
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-04 (Estimated); Study Completion 2029-05-04 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficiency (reference: histopathological diagnosis) | 6 months
  Sensitivity, Specificity, Area under the receiver operation characteristic curve, positive and negative predictive values.

SECONDARY OUTCOMES:
Diagnostic efficiency of ctDNA combined with imaging (ultrasonography, MRI, PET-CT, CT, etc.) and CA 125 for differentiation of benign and malignant adnexal masses. | 6 months
  Area under the receiver operation characteristic curve, sensitivity, specificity, positive and negative predictive values.
Disease stage | 6 months
  FIGO stage
Treatment response | 2 years
  Response to treatment
Survival | 5 years
  Survival rate
Tumour Biology | 6 months
  Mutational profile assessed by Whole Exome Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Ina Marie Dueholm Hjorth, MD, Principal Investigator — University of Aarhus
Locations (1):
- Department of Gynaecology and Obstetrics, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
Depending on GDPR regulations